CLINICAL TRIAL: NCT01573572
Title: A Phase IV, Open Label, Multi-center Study to Assess the Effect of Intravitreal Injections of Macugen (Pegaptanib Sodium Injection) Administered Every 6 Weeks for 48 Weeks on the Corneal Endothelium.
Brief Title: Extension Study to Gather Data on Effect of Macugen on the Corneal Endothelium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EOP 1024
Record Dates: First submitted 2011-02-04; First posted 2012-04-09 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Age-Related Macular Degeneration; Retinal Vein Occlusion; Diabetic Macular Edema
MeSH Terms: conditions — Macular Degeneration; Retinal Vein Occlusion | interventions — pegaptanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravitreal Injections of Macugen (Experimental)
  Interventions: Drug: pegaptanib sodium injection

INTERVENTIONS:
Drug: pegaptanib sodium injection — 0.3mg of Macugen in a single-use, prefilled glass syringe given every 6 weeks for 48 weeks
  Other Names: Macugen

SUMMARY:
This study was conducted because the FDA requested clinical information on potential effects of intravitreal injections of Macugen (pegaptanib sodium injection) on the corneal endothelium from a 1-year (minimum) post-approval clinical study to support that there are no adverse effects on the corneal endothelium following intravitreal injections of Macugen.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of either gender aged > or = to 50 years diagnosed with subfoveal neovascular Age-Related Macular Degeneration, Diabetic Macular Edema, or Retinal Vein Occlusion.
2. Best corrected visual acuity in the study eye between 85 and 20 ETDRS letters or between 20/20 and 20/400 using a Snellen chart.
3. Women must be using two forms of effective contraception, be post-menopausal for at least 12 months prior to study entry, or surgically sterile; if of child-bearing potential, a urine pregnancy test must be performed within 7 days prior to the first injection with a negative result. If the test is positive, a serum test must be done to confirm. The two forms of effective contraception must be implemented during the study and for at least 60 days following the last dose of test medication.
4. Provide written informed consent.
5. Ability to return for all study visits.

Exclusion Criteria:

Subjects will not be eligible for the study if subjects cannot attend all study-required visits, or if any of the following criteria are present

1. Unilateral ocular blunt trauma within one year of enrollment and no greater than 5% difference in central endothelial cell density between the 2 eyes.
2. intraocular surgery (cataract surgery and surgery for glaucoma without tube shunt or mini-shunt) within one year of enrollment.
3. Anterior segment laser surgery (laser trabeculoplasty) performed within one year of enrollment.
4. Glaucoma tube-shunt surgery
5. Previous history of corneal transplant in the study or non-study eye
6. Presence of vitreous macular traction
7. Previous therapeutic radiation in the region of the study eye
8. Any treatment with an investigational agent in the past 30 days for any condition
9. Known serious allergies to the components of pegaptanib sodium formulation

Any of the following underlying diseases including:1. History or evidence of severe cardiac disease(e.g. NYHA Functional Class III or IV - see Appendix 2), clinical or medical history of unstable angina, acute coronary syndrome, myocardial infarction or revascularization within 6 months, ventricular tachyarrhythmias requiring ongoing treatment 7. History or evidence of clinically significant peripheral vascular disease, such as intermittent claudication or prior amputation 8. History or evidence of clinically significant impaired renal or hepatic function 8. Stroke (within 12 months of study entry) 9. Any major surgical procedure within one month of study entry 10. Significant media opacities, including cataract, which might interfere with visual acuity, assessment of toxicity. Subjects should not be entered if there is likelihood that they will require cataract or glaucoma surgery in either eye during the study treatment and follow-up period.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2010-04-22 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Kaur, M.D., Study Director — Valeant Pharmaceuticals NA
Locations (4):
- United States (4):
  - Marietta Eye Clinic, Murrieta, California
  - Wolfe Eye Clinic, Marshalltown, Iowa
  - Associates in Ophthalmology, West Mifflin, Pennsylvania
  - Valley Retina Institute, Harlingen, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravitreal Injections of Macugen
Started | 131
Completed | 103
Not Completed | 28

BASELINE CHARACTERISTICS:
Arm/Group | Intravitreal Injections of Macugen
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 81
  More than one race | 0
  Unknown or Not Reported | 40
Designated eye [Count of Participants; unit: Participants]
  Right eye | 69
  Left eye | 62

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Endothelial Cell Density
Description: The effect on the corneal endothelium will be assessed by specular microscopy, by assessing mean cell density change from baseline. This is to evaluate that there are no adverse effects on the corneal endothelium following intravitreal injections of Macugen.
Time Frame: Baseline, Week 54
Population: Participants with cell density assessments at both baseline and Week 54.
Measure: Mean (Standard Deviation); unit: cells/millimeter squared
Arm/Group | Intravitreal Injections of Macugen
Number analyzed (Participants) | 87
cells/millimeter squared | -35.86 (175.544)

ADVERSE EVENTS:
Time Frame: 54 weeks
Arm/Group | Intravitreal Injections of Macugen
All-Cause Mortality (participants affected / at risk) | 4/131
Serious Adverse Events (participants affected / at risk) | 12/131
Other Adverse Events (participants affected / at risk) | 19/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravitreal Injections of Macugen (N=131)
Cardiac failure congestive (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Chest pain (General disorders) | 2
Blood pressure inadequately controlled (Vascular disorders) | 2
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hypernatraemia (Investigations) | 1
Glaucoma (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Pancreatic carcinoma (Gastrointestinal disorders) | 1
Cerebrovascular accident (Vascular disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravitreal Injections of Macugen (N=131)
Eye pain (Eye disorders) | 10
Conjunctival haemorrhage (Eye disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT01573572/Prot_SAP_000.pdf